CLINICAL TRIAL: NCT05263895
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE-DOSE, CROSSOVER STUDY TO ESTIMATE THE RELATIVE BIOAVAILABILITY OF PF-07321332 FOLLOWING ORAL ADMINISTRATION OF 4 DIFFERENT FORMULATIONS RELATIVE TO THE COMMERCIAL TABLET FORMULATION IN HEALTHY ADULT PARTICIPANTS UNDER FASTED CONDITIONS
Brief Title: Relative Bioavailability Study of 4 Different Formulations of PF-07321332 Relative to the Commercial Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4671008; NCT05263895 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-02-25; First posted 2022-03-03 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Bioavailability
Keywords: coronavirus disease 2019 (COVID-19); severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination; nirmatrelvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A: PF-0732133/ritonavir (Active Comparator): PF-07321332 ritonavir
  Interventions: Drug: PF-07321332/ritonavir
- Treatment B: PF-07321332/ritonavir (Experimental): PF-07321332 ritonavir
  Interventions: Drug: PF-07321332/ritonavir
- Treatment C: PF-07321332/ritonavir (Experimental): PF-07321332 ritonavir
  Interventions: Drug: PF-07321332/ritonavir
- Treatment D: PF-07321332/ritonavir (Experimental): PF-07321332 ritonavir
  Interventions: Drug: PF-07321332/ritonavir
- Treatment E: PF-07321332 (Experimental): PF-07321332
  Interventions: Drug: PF-07321332

INTERVENTIONS:
Drug: PF-07321332/ritonavir — PF-07321332 ritonavir will be administered as single dose orally
  Arms: Treatment A: PF-0732133/ritonavir
Drug: PF-07321332/ritonavir — PF-07321332 ritonavir will be administered as single oral dose orally.
  Arms: Treatment B: PF-07321332/ritonavir
Drug: PF-07321332/ritonavir — PF-07321332 ritonavir will be administered as single oral dose orally.
  Arms: Treatment C: PF-07321332/ritonavir
Drug: PF-07321332/ritonavir — PF-07321332 ritonavir will be administered as single oral dose orally.
  Arms: Treatment D: PF-07321332/ritonavir
Drug: PF-07321332 — PF-07321332 will be administered as single oral dose orally.
  Arms: Treatment E: PF-07321332

SUMMARY:
The purpose of this study is to estimate the relative bioavailability of PF-07321332 in different formulations in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination (PE), laboratory tests, vital signs and standard 12 lead ECGs.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures

Exclusion Criteria:

* Positive test result for SARS-CoV-2 infection at the time of Screening or Day -1.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinically relevant abnormalities requiring treatment (eg, acute myocardial infarction, unstable ischemic conditions, evidence of ventricular dysfunction, serious tachy or brady arrhythmias) or indicating serious underlying heart disease (eg, prolonged PR interval, cardiomyopathy, heart failure greater than New York Heart Association (NYHA) 1, underlying structural heart disease, Wolff Parkinson-White syndrome).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis B surface antibody (HCVAb). Hepatitis B vaccination is allowed.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
* Participant who have received a COVID-19 vaccine within 7 days before screening or admission, or who are to be vaccinated with a COVID-19 vaccine at any time during the study confinement period.
* A positive urine drug test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Sagawa K, Lin J, Jaini R, Di L. Physiologically-Based Pharmacokinetic Modeling of PAXLOVID with First-Order Absorption Kinetics. Pharm Res. 2023 Aug;40(8):1927-1938. doi: 10.1007/s11095-023-03538-5. Epub 2023 May 25. PMID 37231296
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671008

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twelve participants were enrolled to 1 of 6 sequences. Each participant participated in 5 study periods to receive 5 treatments: Treatment A: nirmatrelvir (commercial tablets)/ritonavir 300/100 mg; Treatment B: nirmatrelvir (slower dissolution tablets)/ritonavir 300/100 mg; Treatment C: nirmatrelvir (large particle size tablets)/ritonavir 300/100 mg; Treatment D: nirmatrelvir (spray dried dispersion [SDD] suspension)/ritonavir 300/100 mg; Treatment E: nirmatrelvir 300 mg (SDD suspension)
Groups:
- Sequence 1: Twelve participants were randomly assigned to 1 of 6 sequences. Each sequence included 2 participants who received 5 study treatments in 5 study periods.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg commercial tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 1.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg slower dissolution tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 2.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg larger particle size tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 3.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 4.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally without ritonavir starting at approximately 0800 hours (plus or minus 2 hours) in Period 5.
- Sequence 2: On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg slower dissolution tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 1.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg larger particle size tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 2.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg commercial tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 3.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 4.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally without ritonavir starting at approximately 0800 hours (plus or minus 2 hours) in Period 5.
- Sequence 3: On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg larger particle size tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 1.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg commercial tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 2.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg slower dissolution tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 3.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 4.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally without ritonavir starting at approximately 0800 hours (plus or minus 2 hours) in Period 5.
- Sequence 4: On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg commercial tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 1.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg larger particle size tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 2.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg slower dissolution tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 3.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally without ritonavir starting at approximately 0800 hours (plus or minus 2 hours) in Period 4.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 5.
- Sequence 5: On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg slower dissolution tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 1.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg commercial tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 2.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg larger particle size tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 3.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally without ritonavir starting at approximately 0800 hours (plus or minus 2 hours) in Period 4.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 5.
- Sequence 6: On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg larger particle size tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 1.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg slower dissolution tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 2.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg commercial tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 3.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally without ritonavir starting at approximately 0800 hours (plus or minus 2 hours) in Period 4.
  On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours) in Period 5.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who took at least 1 dose of study intervention.
Groups:
- All Participants: All participants enrolled in this study, "Enrolled" meant a participant's agreement to participate in a clinical study following completion of the informed consent process and screening. Potential participants who were screened for the purpose of determining eligibility for the study, but did not participate in the study, were not considered enrolled, unless otherwise specified by the protocol. A participant was considered enrolled if the informed consent was not withdrawn prior to participating in any study activity after screening.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: Years] | 48.0 [35 to 62]
Age, Customized [Number; unit: Participants]
  <18 years | 0
  18-44 years | 5
  45-64 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 6
    Black or African American | 5
    Black or African American, White | 1
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 11

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (Clast) (AUClast) of Nirmatrelvir
Description: AUClast for nirmatrelvir was calculated by Linear/Log trapezoidal method. Natural log-transformed AUClast for nirmatrelvir (slower dissolution tablets and large particle size tablets) was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Natural log-transformed AUClast for Nirmatrelvir (SDD suspension) was analyzed using a mixed effect model with sequence and treatment as fixed effects and participant within sequence as a random effect.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours postdose
Population: All participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg: On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg commercial tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours).
- Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg: On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg slower dissolution tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours).
- Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg: On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as 2 × 150 mg larger particle size tablets, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours).
- Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg: On Day 1, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally with ritonavir 100 mg (as 1 × 100 mg tablet) starting at approximately 0800 hours (plus or minus 2 hours).
- Nirmatrelvir (SDD Suspension) 300 mg: On Day, following an overnight fast of at least 10 hours, participants received nirmatrelvir 300 mg as SDD suspension, administered orally without ritonavir starting at approximately 0800 hours (plus or minus 2 hours).
Arm/Group | Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension) 300 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 35020 (15) | 31700 (26) | 35990 (26) | 48380 (15) | 10530 (50)
Statistical Analysis 1: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg; Test: Nirmatrelvir (slower dissolution tablets)/ritonavir 300/100 mg Reference: Nirmatrelvir (commercial tablets)/ritonavir 300/100 mg; Test type: Other; Ratio of Adjusted Geometric means = 90.54, 90% CI 2-sided [79.85 to 102.65]
Statistical Analysis 2: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg; Test: Nirmatrelvir (large particle size tablets)/ritonavir 300/100 mg Reference: Nirmatrelvir (commercial tablets)/ritonavir 300/100 mg; Test type: Other; Ratio of Adjusted Geometric Means = 102.78, 90% CI 2-sided [90.65 to 116.53]
Statistical Analysis 3: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg; Test: Nirmatrelvir (SDD suspension)/ritonavir 300/100 mg Reference: Nirmatrelvir (commercial tablets)/ritonavir 300/100 mg; Test type: Other; Ratio of Adjusted Geometric Means = 138.15, 90% CI 2-sided [118.03 to 161.69]
Statistical Analysis 4: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (SDD Suspension) 300 mg; Test: Nirmatrelvir (SDD suspension) 300 mg Reference: Nirmatrelvir (commercial tablets)/ritonavir 300/100 mg; Test type: Other; Ratio of Adjusted Geometric Means = 30.8, 90% CI 2-sided [25.70 to 35.20]

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of Nirmatrelvir
Description: AUCinf for nirmatrelvir was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve. Natural log-transformed AUCinf for nirmatrelvir (slower dissolution tablets and large particle size tablets) was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Natural log-transformed AUCinf for Nirmatrelvir (SDD suspension) was analyzed using a mixed effect model with sequence and treatment as fixed effects and participant within sequence as a random effect.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension) 300 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng*hr/mL | 35540 (14) | 32430 (26) | 36420 (25) | 48680 (15) | 10580 (50)
Statistical Analysis 1: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 91.26, 90% CI 2-sided [80.46 to 103.51]
Statistical Analysis 2: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 102.49, 90% CI 2-sided [90.36 to 116.26]
Statistical Analysis 3: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg; [analysis description as in outcome 1, analysis 3]; Test type: Other; Ratio of Adjusted Geometric Means = 136.99, 90% CI 2-sided [117.09 to 160.27]
Statistical Analysis 4: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (SDD Suspension) 300 mg; Test: Nirmatrelvir (SDD suspension) 300 mg Reference: Nirmatrelvir (commercial tablets)/ritonavir 300/100 mg; Test type: Other; Ratio of Adjusted Geometric Means = 29.77, 90% CI 2-sided [25.45 to 34.83]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Nirmatrelvir
Description: Cmax for nirmatrelvir was observed directly from data. Natural log-transformed Cmax for nirmatrelvir (slower dissolution tablets and large particle size tablets) was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Natural log-transformed Cmax for Nirmatrelvir (SDD suspension) was analyzed using a mixed effect model with sequence and treatment as fixed effects and participant within sequence as a random effect.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension) 300 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng/mL | 3347 (16) | 3155 (23) | 3635 (27) | 8840 (14) | 4871 (30)
Statistical Analysis 1: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 94.28, 90% CI 2-sided [80.77 to 110.05]
Statistical Analysis 2: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 108.60, 90% CI 2-sided [93.04 to 126.76]
Statistical Analysis 3: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg; [analysis description as in outcome 1, analysis 3]; Test type: Other; Ratio of Adjusted Geometric Means = 264.12, 90% CI 2-sided [232.32 to 300.27]
Statistical Analysis 4: Comparison: Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg vs Nirmatrelvir (SDD Suspension) 300 mg; Test: Nirmatrelvir (SDD suspension) 300 mg Reference: Nirmatrelvir (commercial tablets)/ritonavir 300/100 mg; Test type: Other; Ratio of Adjusted Geometric Means = 145.53, 90% CI 2-sided [128.01 to 165.45]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs might arise from symptoms or other complaints reported to the investigator by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative), or they might arise from clinical findings of the investigator or other healthcare providers (clinical signs, test results, etc.). TEAEs were those with initial onset or increasing in severity after the first dose of study treatment.
Time Frame: Baseline up to 35 days after last dose of study intervention (up to 12 weeks)
Population: All participants who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension) 300 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants
  All-Causality AEs | 4 | 1 | 3 | 0 | 1
  Treatment-Related AEs | 4 | 1 | 1 | 0 | 1

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: The laboratory abnormality parameters included Chemistry: bicarbonate (milliequivalents per liter [mEq/L]) <0.9 x lower limit of normal (LLN), urobilinogen (ehrlich units per deciliter [EU/dL]) >=1, and fibrinogen (milligram/deciliter [mg/dL]) >1.25 x baseline; Urinalysis: URINE hemoglobin (Scalar) >=1, only those categories in which at least 1 participant had data were reported. All the safety laboratory samples were collected following at least a 4 hour fast. Clinical laboratory evaluations only included treatments of nirmatrelvir SDD suspension/ritonavir 300/100 mg and nirmatrelvir SDD suspension 300 mg. No participant was evaluable for clinical laboratory evaluations for the other treatments.
Time Frame: Screening (from Day-28 to Day-2), Day-1 of Period 1 (before 1st dose) and Day4 of Period 5 (4 days after the last dose on study discharge day). Each treatment period was 4 days long (Day1 to Day4) with a minimum of 4 days washout between each period
Population: Participants with at least 1 observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension) 300 mg
Number analyzed (Participants) | 6 | 6
Participants
  Bicarbonate (mEq/L) <0.9 x LLN | 1 | 0
  Urobilinogen (EU/dL) >=1 | 1 | 0
  Fibrinogen (mg/dL) >1.25 x Baseline | 0 | 1
  URINE Hemoglobin (Scalar) >=1 | 1 | 0

6. Secondary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Single supine blood pressure (BP) and pulse rate (PR) were measured with the participant's arm supported at the level of the heart and recorded to the nearest mm Hg after approximately 5 minutes of rest. The same arm (preferably the dominant arm) was used throughout the study. Participants were instructed not to speak during measurements.
Time Frame: Screening (D28-D2), D1 of Period 1 (before 1st dose), D1 hr 0,2,and 6 of each period, and D4 of Period 5 (4 days after the last dose on study discharge day). Each treatment Period was 4 days long (D1-D4) with a minimum 4 days washout between each period
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension) 300 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With ECG Abnormalities
Description: Standard 12-lead ECGs utilizing limb leads (with a 10 second rhythm strip) were collected. All scheduled ECGs were performed after the participant had rested quietly for at least 5 minutes in a supine position.
Time Frame: Screening (from D-28 to D-2), D1, hr0 of Period 1 (before 1st dose) and D4 of Period 5 (4 days after last dose on study discharge day). Each treatment period was 4 days long (D1 to D4) with a minimum of 4 days washout between each period
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension) 300 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Physical Examination Abnormalities
Description: A complete PE included, at a minimum, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, and gastrointestinal, musculoskeletal, and neurological systems. A brief physical examination included, at a minimum, assessments of general appearance, the respiratory and cardiovascular systems, and participant reported symptoms.
Time Frame: Screening (from Day-28 to Day-2), Day-1 of Period 1 (before 1st dose. Each treatment period was 4 days long (Day1 to Day4) with a minimum of 4 days washout between each period
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension) 300 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 35 days after last dose of study intervention (up to 12 weeks)
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg | Nirmatrelvir (SDD Suspension) 300 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 1/12 | 3/12 | 0/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nirmatrelvir (Commercial Tablets)/Ritonavir 300/100 mg (N=12) | Nirmatrelvir (Slower Dissolution Tablets)/Ritonavir 300/100 mg (N=12) | Nirmatrelvir (Large Particle Size Tablets)/Ritonavir 300/100 mg (N=12) | Nirmatrelvir (SDD Suspension)/Ritonavir 300/100 mg (N=12) | Nirmatrelvir (SDD Suspension) 300 mg (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT05263895/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT05263895/SAP_001.pdf